CLINICAL TRIAL: NCT05203614
Title: Positive Activities for Asian American Cancer Patients and Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-0998; NCI-2021-12848 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2021-11-11; First posted 2022-01-24 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Household Contribution (Other): Do something thoughtful or nice for your caregiver that would provide them with tangible support
  Interventions: Behavioral: Household Contribution
- Outside Contribution (Other): Do something outside your home/household that contributes to the larger society
  Interventions: Behavioral: Outside Contribution
- Control (Other): Keep track of your daily activities
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Household Contribution — Questionnaires
  Arms: Household Contribution
Behavioral: Outside Contribution — Questionnaires
  Arms: Outside Contribution
Behavioral: Control — Questionnaires
  Arms: Control

SUMMARY:
Positive Activities for Asian American Cancer Patients and Caregivers

DETAILED DESCRIPTION:
Primary Objectives:

The overall objective of this project is to design and test the feasibility of two positive activities, household contribution and outside contribution, to increase quality of life in AA cancer patients.

Secondary Objectives:

Aim 1: To assess the acceptability and feasibility of household and outside contribution positive activities for AAs through a mixed qualitative and exploratory quantitative investigation.

Aim 2: To use the qualitative and quantitative data from Aim 1, in collaboration with the mentorship team, AA community members, and clinicians, to develop one or both positive activity intervention(s) (i.e., household or outside contribution) specifically for AA cancer patients.

ELIGIBILITY:
Inclusion criteria for patients will be:

* self-identifies as AA,
* males or females ages 25-75 years
* within 1 year of any cancer diagnosis
* actively undergoing systemic therapy (e.g., chemotherapy, radiation)
* able to identify a caregiver (e.g., spouse) who lives in the same household and consents to participate in the study,
* able to read, write, and speak English (i.e., English proficient; EP),
* access to internet, computer/phone, and web browser.

Exclusion criteria for patients will be:

* life expectancy less than 6 months in the opinion of the primary physician,
* inability to stand or walk on their own or other physical limitations that preclude them from participating (3+ on ECOG performance status),
* major thought disorder (e.g., schizophrenia or bipolar [patient records or

Inclusion criteria for caregivers will be:

* identifies as AA,
* patient considers them to be caregiver, -
* EP,
* access to computer/phone, internet, and web browser.

Exclusion criteria for caregivers will be:

* unwilling or unable to participate in the study for any reason,
* under the age of 18.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Quality of Life Questionnaires(HRQOL & interpersonal well-being ) | through study completion, an average of 1 year
  Hedonic well-being (positive and negative emotions) will be measured using a modified 12-item Affect-Adjective Scale (AAS)42 that includes low-arousal emotion items (e.g., peaceful/serene, dull/bored).

CONTACTS AND LOCATIONS:
Overall Officials: LI Qian, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-11-11): https://cdn.clinicaltrials.gov/large-docs/14/NCT05203614/ICF_000.pdf